CLINICAL TRIAL: NCT03784625
Title: Targeted Radionuclide Therapy for Metastatic Melanoma [131I] ICF01012: Phase I Study
Brief Title: Targeted Radionuclide Therapy for Metastatic Melanoma [131I] ICF01012
Acronym: MELRIV-1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002444-17; TRANSLA12-143 (Other Grant/Funding Number: Ministry of Health, National Cancer Institute, France)
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
Keywords: metastatic melanoma; targeted radionuclide therapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: dose escalation model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- therapeutic dose activity (level 1) (Experimental): [131]ICF01012 at a therapeutic dose of 800 MBq/m² , single dose at D11 (intravenous administration)
  Interventions: Drug: [131I]ICF01012 (therapeutic dose level 1)
- therapeutic dose activity (level 2) (Experimental): [131]ICF01012 at a therapeutic dose of 1600 MBq/m² , single dose at D11 (intravenous administration)
  Interventions: Drug: [131I]ICF01012 (therapeutic dose level 2)
- therapeutic dose activity (level 3) (Experimental): [131]ICF01012 at a therapeutic dose of 2700 MBq/m² , single dose at D11 (intravenous administration)
  Interventions: Drug: [131I]ICF01012 (therapeutic dose level 3)
- therapeutic dose activity (level 4) (Experimental): [131]ICF01012 at a therapeutic dose of 4000 MBq/m² , single dose at D11 (intravenous administration)
  Interventions: Drug: [131I]ICF01012 (therapeutic dose level 4)

INTERVENTIONS:
Drug: [131I]ICF01012 (therapeutic dose level 1) — * 1 diagnostic injection (D0) at a diagnostic dose of 185 MBq. This first dose permits to pre-select patients who will received a therapeutic dose according to the dosimetry results ( binding on at least a tumoral lesion, an acceptable radiation absorbed dose to major organs)
  * 1 therapeutic injection (D11) at a dose of 800 MBq/m²
  Arms: therapeutic dose activity (level 1)
Drug: [131I]ICF01012 (therapeutic dose level 2) — * 1 diagnostic injection (D0) at a diagnostic dose of 185 MBq. This first dose permits to pre-select patients who will received a therapeutic dose according to the dosimetry results ( binding on at least a tumoral lesion, an acceptable radiation absorbed dose to major organs)
  * 1 therapeutic injection (D11) at a dose of 1600 MBq/m²
  Arms: therapeutic dose activity (level 2)
Drug: [131I]ICF01012 (therapeutic dose level 3) — * 1 diagnostic injection (D0) at a diagnostic dose of 185 MBq. This first dose permits to pre-select patients who will received a therapeutic dose according to the dosimetry results ( binding on at least a tumoral lesion, and an acceptable radiation absorbed dose to major organs)
  * 1 therapeutic injection (D11) at a dose of 2700 MBq/m²
  Arms: therapeutic dose activity (level 3)
Drug: [131I]ICF01012 (therapeutic dose level 4) — * 1 diagnostic injection (D0) at a diagnostic dose of 185 MBq. This first dose permits to pre-select patients who will received a therapeutic dose according to the dosimetry results ( binding on at least a tumoral lesion, and an acceptable radiation absorbed dose to major organs)
  * 1 therapeutic injection (D11) at a dose of 4000 MBq/m²
  Arms: therapeutic dose activity (level 4)

SUMMARY:
This study is a phase I clinical trial aimed to determine the recommended dose of [131I]ICF01012 to administer for the treatment of patients with pigmented metastatic melanoma (binding [131I]ICF01012 ). The [131I]ICF01012 is a targeted radionuclide therapy with a high affinity for melanin.

DETAILED DESCRIPTION:
This study will include a maximum of 36 patients. This study will begin with a preselection part that consists of an injection of [131I]ICF01012 at a diagnostic dose (185 MBq) in order to preselect patients who will receive the therapeutic dose according to the dosimetry results : binding of [131I]ICF01012 on at least a tumoral lesion and an acceptable radiation absorbed dose to major organs.

The second phase will consist of a therapeutic part with a single administration of [131I]ICF01012 at a therapeutic dose. This part is a dose escalation model (4 levels of therapeutic dose were tested)

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic melanoma failure to recommended treatments by HAS.
* Initial histological diagnosis of cutaneous melanoma pigmented or unknown status or choroidal melanoma.
* Presence of at least one measurable lesion and / or evaluable in 18FDG-PET as PERCIST criteria.
* Presence of at least one measurable lesion and / or evaluable as CT RECIST 1.1 criteria.
* WHO performance index ≤ 2 .
* Age> 18 years
* Life expectancy> 3 months.
* Creatinine ≤ 1,5 x ULN or creatinine clearance ≥ 60ml/min if creatinine > 1,5 x ULN , Neutrophil > 1,5.109L-1, Platellets > 100 x 109L-1, prothrombine time < 1,3 x control, Hemoglobin > 9 g/dL, facteur V > 80% (or AST, ALT ≤ 3 x LNS (≤ 5 x ULN if liver metastasis)).
* Normal cardiac fonction (LVEF> 40%).

Exclusion Criteria:

* Brain metastases symptomatic
* Patient with a VI skin phototype
* Previous treatment with chemotherapy, radiotherapy, immunotherapy and targeted therapy in the previous 4 weeks, the first injection of [131I] ICF01012
* Pregnant woman, nursing or woman of childbearing age refusing to follow effective contraception during treatment and 12 months after the administration of therapeutic dose.
* Men refusing to follow effective contraception during treatment and 12 months after the administration of therapeutic dose
* Other evolutionary known cancer in the past five years
* Earlier irradiation of more than 25% of the bone marrow
* Suspicion of invasion of more than 25% of the bone marrow on imaging 18F-FDG PET-CT
* External Radiotherapy on target organs or the maximum dose as recommended in force
* Uncontrolled diabetes
* Known history of allergy to the excipients of the solution of [131I]ICF01012
* Any comorbidity or severe disease at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of the recommended therapeutic dose of [131I] ICF01012 | Only toxicities observed during the 6 weeks following administration of the therapeutic dose will be considered for the evaluation of DLT
  defined as the highest dose at which the percentage of DLT (dose limiting toxicity) is less than 33%. The DLT is defined as:
  * all non hematologic toxicities NCI-CTC grade 3-4 except for alopecia, nausea, vomiting and fever that can be controlled by appropriate measures.
  * hematologic toxicities as thrombopenia and anemia of grade 4, neutropenia of grade 4 for more than 5 days, thrombopenia of grade 3 with bleeding and all other hematologic toxicities of grade 3 clinically significant of more than 3 weeks

SECONDARY OUTCOMES:
Evaluation of the sensitivity and specificity by patients and by lesions of [131I]ICF01012 ICF01012 for the visualization of metastatic melanoma lesions from the examinations made during the selection phase | selection phase Day 0 - Day 7
  binding of [131I]ICF01012 compared to standard evaluation of metastatic lesion (standard imaging (CT Scan, TEP ...) or clinical evaluation)
Evaluation of the tolerance of [131I] ICF01012 (adverse events assessed by NCI-CTC Version 4.03) | from the the first dose to the end of study (3 months after diagnostic dose)
  adverse events assessed by NCI-CTC Version 4.03
Pharmacokinetics of [131I] ICF01012 including the study of biodistribution and excretion (radiation counting of serum, whole blood and urinary samples) | selection phase Day 0 (diagnostic dose), Day 1, and Day 4, Day 7
  radiation counting of serum, whole blood and urinary samples
Evaluation of the therapeutic response of [131I] ICF01012. | at 3 months
  Response will be categorized according to the criteria from RECIST 1.1 and PERCIST criteria: complete response, partial response, stable disease and progressive disease
Evaluation of personal dosimetry for the administration of [131I]ICF01012. | Selection phase : Day 0, Day 1, Day 4, and Day 7; therapeutic phase : Day 15, Day 18 and Day 25, Day 74
  assessed by whole-body planar studies and tomographic imaging with single-photon emission computed tomography (SPECT)/CT

CONTACTS AND LOCATIONS:
Overall Officials: Florent CACHIN, Pr, Principal Investigator — Centre Jean Perrin
Locations (2):
- France (2):
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Clermont-Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thivat E, Rouanet J, Auzeloux P, Sas N, Jouberton E, Levesque S, Billoux T, Mansard S, Molnar I, Chanchou M, Fois G, Maigne L, Chezal JM, Miot-Noirault E, D'Incan M, Durando X, Cachin F. Phase I study of [131I] ICF01012, a targeted radionuclide therapy, in metastatic melanoma: MELRIV-1 protocol. BMC Cancer. 2022 Apr 15;22(1):417. doi: 10.1186/s12885-022-09495-3. PMID 35428211